CLINICAL TRIAL: NCT03356938
Title: The Role of the Circadian System in Neurological Sleep-wake Disorders: Assessment of Circadian and Homeostatic Sleep-wake Regulation and Vigilance With a Poly-nap Protocol
Brief Title: The Role of the Circadian System in Neurological Sleep-wake Disorders
Acronym: PNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esther Werth (Other)
Responsible Party: Sponsor-Investigator, Esther Werth, Head of Sleep Laboratory, University of Zurich
Organization: University of Zurich (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHPNP2016
Record Dates: First submitted 2017-11-15; First posted 2017-11-29 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Narcolepsy 1; Idiopathic Hypersomnia
MeSH Terms: conditions — Narcolepsy 1; Idiopathic Hypersomnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline recording (No Intervention)
- Sleep restriction (Experimental)
  Interventions: Behavioral: Sleep restriction
- Sleep deprivation (Experimental)
  Interventions: Behavioral: Sleep deprivation

INTERVENTIONS:
Behavioral: Sleep restriction — Restricted sleep to 5 hours / night for 5 days prior to sleep laboratory examination
  Arms: Sleep restriction
Behavioral: Sleep deprivation — Sleep deprivation during first night of sleep laboratory examination
  Arms: Sleep deprivation

SUMMARY:
The aim of this study is to investigate the role of the circadian system in patients with neurologic sleep-wake disorders. Therefore, overnight sleep will be distributed over 30 hours into repetitive sleep-wake cycles (poly-nap protocol), so that sleep episodes occur at different circadian phases. Vigilance, attention, risk behavior as well as sleep onset latency will be observed.

Ambulatory accelerometer recordings gain more and more attention in the diagnostic work-up of sleep disorders, as they allow to also include the everyday rest-activity rhythm before examinations in the sleep laboratory. Advances of novel devices should improve the detection of rest and activity and therefore the estimation of sleep and wake, especially in patients with neurologic sleep-wake disorders exhibiting fragmented sleep. Two types of actimeters will be applied throughout our study protocol to explore better classification of sleep and wake phases and patterns of the rest-activity rhythm.

This study is designed as an observational case-controlled study targeting the disorders of narcolepsy type 1 and idiopathic hypersomnia, and including interventional procedures in the healthy control group (sleep deprivation, sleep restriction) in a counter-balanced design.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female participants 18 years to 35 years of age
* Written informed consent by the participant after information about the research project
* Healthy controls: 7-8 hours of sleep per night
* Healthy controls: sleep satiation before start of the study
* Narcolepsy type 1: diagnosis of narcolepsy with cataplexy, drug free during study, proven excessive daytime sleepiness with increased REM (MSLT), clear-cut cataplexy present, undetectable or low cerebrospinal fluid hypocretin levels (if data is available)
* Idiopathic hypersomnia: diagnosis of idiopathic hypersomnia, drug free during study, proven excessive daytime sleepiness without increased REM (MSLT), increased sleep need (>10h/day) on work-free days shown by 2-week actigraphy

Exclusion Criteria:

* signs of neurological, psychiatric, or other sleep-wake disorders
* signs of sleep deprivation
* shift work and time zone change of more than one hour within one month prior the study start
* extreme morning and evening types
* underweight
* obstructive gastro-intestinal disease or history of gastrointestinal surgery
* an implanted medical device or a scheduled MRI scan during the experimental period

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Endogenous melatonin | Half an hour before and half an hour after a nap during PNP protocol, up to 2 minutes.
  Dim light melatonin onset (DLMO) will show whether there is a phase difference between patient groups and between patients and controls. The amplitude of the melatonin profile will show whether there is a dampening of the circadian rhythm or not.
EEG slow-wave activity (SWA) | Over nap times, up to 80 minutes.
  SWA is a marker of homeostatic sleep pressure and will show whether patients with narcolepsy or idiopathic hypersomnia live under different sleep pressure than controls.

SECONDARY OUTCOMES:
Performance in neurobehavioral tests | One hour before each nap, up to 45mins.
  Outcome for vigilance and cognition of the subjects.
EEG event related potentials (ERPs) | One hour before each nap, up to 45minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Werth, PhD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borbely AA. A two process model of sleep regulation. Hum Neurobiol. 1982;1(3):195-204. No abstract available. PMID 7185792
- [Background] Dauvilliers Y, Arnulf I, Mignot E. Narcolepsy with cataplexy. Lancet. 2007 Feb 10;369(9560):499-511. doi: 10.1016/S0140-6736(07)60237-2. PMID 17292770
- [Background] Frenette E, Kushida CA. Primary hypersomnias of central origin. Semin Neurol. 2009 Sep;29(4):354-67. doi: 10.1055/s-0029-1237114. Epub 2009 Sep 9. PMID 19742411
- [Background] Munch M, Knoblauch V, Blatter K, Schroder C, Schnitzler C, Krauchi K, Wirz-Justice A, Cajochen C. Age-related attenuation of the evening circadian arousal signal in humans. Neurobiol Aging. 2005 Oct;26(9):1307-19. doi: 10.1016/j.neurobiolaging.2005.03.004. Epub 2005 Apr 18. PMID 16182904
- [Background] Saper CB, Scammell TE, Lu J. Hypothalamic regulation of sleep and circadian rhythms. Nature. 2005 Oct 27;437(7063):1257-63. doi: 10.1038/nature04284. PMID 16251950
- [Background] Wulff K, Gatti S, Wettstein JG, Foster RG. Sleep and circadian rhythm disruption in psychiatric and neurodegenerative disease. Nat Rev Neurosci. 2010 Aug;11(8):589-99. doi: 10.1038/nrn2868. Epub 2010 Jul 14. PMID 20631712
- [Background] Morgenthaler T, Alessi C, Friedman L, Owens J, Kapur V, Boehlecke B, Brown T, Chesson A Jr, Coleman J, Lee-Chiong T, Pancer J, Swick TJ; Standards of Practice Committee; American Academy of Sleep Medicine. Practice parameters for the use of actigraphy in the assessment of sleep and sleep disorders: an update for 2007. Sleep. 2007 Apr;30(4):519-29. doi: 10.1093/sleep/30.4.519. PMID 17520797
- [Derived] Ryser F, Gassert R, Werth E, Lambercy O. A novel method to increase specificity of sleep-wake classifiers based on wrist-worn actigraphy. Chronobiol Int. 2023 May;40(5):557-568. doi: 10.1080/07420528.2023.2188096. Epub 2023 Mar 20. PMID 36938627